CLINICAL TRIAL: NCT00614328
Title: Feasibility and Tolerability of a Combination of Naltrexone and Baclofen for Alcohol Dependence: A Pilot Study.
Brief Title: Combination of Naltrexone and Baclofen for Alcohol Dependence:A Pilot Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: James C. Garbutt, M.D., Principal Investigator, UNC-Chapel Hill, Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 05-2988 GCRC 2497; IRB#05-2988
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol; Alcohol Abuse; Alcohol Drinking
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Naltrexone; Baclofen; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Naltrexone (50 mg once a day) + placebo baclofen + behavioral therapy (n=10)
  Interventions: Drug: Naltrexone, Baclofen, Placebo and Behavior Therapy
- 2 (Active Comparator): Placebo naltrexone + baclofen (10 mg t.i.d) + behavior therapy (n=10)
  Interventions: Drug: Naltrexone, Baclofen, Placebo and Behavior Therapy
- 3 (Active Comparator): Baclofen (10 mg t.i.d) + naltrexone (50 mg once per day) + behavior therapy (n=10)
  Interventions: Drug: Naltrexone, Baclofen, Placebo and Behavior Therapy
- 4 (Placebo Comparator): Placebo baclofen + placebo naltrexone + behavior therapy
  Interventions: Drug: Naltrexone, Baclofen, Placebo and Behavior Therapy

INTERVENTIONS:
Drug: Naltrexone, Baclofen, Placebo and Behavior Therapy — Naltrexone 50mg/day for 12 weeks Baclofen 10mg tid = 30mg/day for 12 weeks Behavior Therapy 9 sessions
  Other Names: Naltrexone/ ReVia

SUMMARY:
The purpose of this research study is to learn about the use of a combination of two medications, baclofen and naltrexone, for the treatment of alcohol dependence in men and women ages 25-60 years old. Naltrexone is an FDA approved medication for treatment of alcohol dependence. The most widely accepted idea for naltrexone's effect is that it reduces the alcohol "high", which decreases a desire to consume alcohol. As a result, alcoholic patients treated with naltrexone are less likely to relapse to heavy drinking. Furthermore, naltrexone treated patients drink fewer days and are more likely to maintain abstinence.

However, naltrexone does not have any effect on other symptoms that may contribute to relapse such as anxiety, sleep problems and irritability. Baclofen, an FDA approved medication for muscle spasms, may improve some of these symptoms.

Therefore, the purpose of the current study is to gather information on whether adding baclofen to naltrexone is feasible and well tolerated.

DETAILED DESCRIPTION:
The purpose of this research study is to learn about the use of a combination of two medications, baclofen and naltrexone, for the treatment of alcohol dependence in men and women ages 25-60 years old. Naltrexone is an FDA approved medication for treatment of alcohol dependence. The most widely accepted idea for naltrexone's effect is that it reduces the alcohol "high", which decreases a desire to consume alcohol. As a result, alcoholic patients treated with naltrexone are less likely to relapse to heavy drinking. Furthermore, naltrexone treated patients drink fewer days and are more likely to maintain abstinence.

However, naltrexone does not have any effect on other symptoms that may contribute to relapse such as anxiety, sleep problems and irritability. Baclofen, an FDA approved medication for muscle spasms, may improve some of these symptoms.

Baclofen has been studied for alcoholism in Italy in 45 individuals in two studies. In the two Italian studies, baclofen significantly reduced alcohol withdrawal symptoms and craving for alcohol, as well as the use of alcohol. These data have been supported by the results of our own pilot study conducted here at UNC in 12 subjects with alcohol dependence. That study showed that baclofen was generally well tolerated, and some individuals had significant improvements in their drinking. Furthermore, we have recently completed enrolling 80 alcohol dependent patients into a placebo-controlled study of baclofen and are currently analyzing the data.

Therefore, the purpose of the current study is to gather information on whether adding baclofen to naltrexone is feasible and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Forty men and women between the ages of 25 to 60 years meeting DSM-IV criteria for current alcohol dependence.
2. Subjects must either have been admitted to UNC Hospitals for a medical detoxification from alcohol and be receiving benzodiazepines for detoxification or recruited from the general population.
3. Must have had at least 2 heavy drinking days (≥5 drinks/day for men or ≥4 drinks/day for women) per week, on average and an average overall consumption of 21 drinks/week or more for men and 14 drinks/week or more for women during the 4 weeks prior to admission or screening and no more than three months of abstinence in the previous year.
4. Able to understand and sign written informed consent.
5. Willingness to engage in treatment and motivation to achieve abstinence or to greatly reduce alcohol consumption.
6. Must have a stable residence and be able to identify an individual who could locate subject if needed.
7. Must have the logistical ability to come to study visits.(This study is being conducted in Chapel Hill, NC. Therefore participants must be able to attend each clinic visit for 12 weeks.)

Exclusion Criteria:

1. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., cirrhosis, kidney impairment, unstable hypertension, hypotension, diabetes mellitus, seizure disorder).
2. Patients taking glucocorticoids or immunosuppressants.
3. Clinically significant psychiatric illness including any psychotic disorder, bipolar disorder, severe depression, persistent suicidal ideation or suicide attempt, or substance use dependence other than alcohol or nicotine.
4. Any prior history of, or currently presenting with, withdrawal seizure or delirium tremens.
5. AST, or ALT > 3 times Upper Limit of Normal (ULN), or bilirubin > ULN, or estimated glomerular filtration rate < 60.
6. Positive urine toxicology screen with the exception of cannabis or cocaine for inpatients only. Patients recruited from the general population who present with a positive urine toxicology screen other than cannabis will be excluded. Any subject with positive cannabis or cocaine screens will be excluded if they have a history of dependence.
7. Concurrent use of mood stabilizers, antipsychotics, stimulants, or hypnotics. Use of benzodiazepines is prohibited except during the withdrawal period for inpatients. Antidepressant medication is permitted.
8. Concurrent use of anticonvulsants, insulin, or oral hypoglycemics.
9. Concurrent use of opiates or any use of opiates within 7 days prior to Naltrexone use.
10. Participation in any clinical trial within the last 60 days.
11. Court-mandated participation in alcohol treatment or pending incarceration.
12. For inpatients, lack of urine toxicology or pregnancy test done on date of hospital admission. Outpatient subjects will have a urine toxicology screen and a pregnancy test done (if female).
13. If female, pregnant or breastfeeding women and women of child bearing potential who do not practice a medically acceptable form of birth control.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
This is an exploratory study to gain experience with the combination of baclofen+naltrexone and to gather pilot data on cytokine levels. Initial interest is in recruitment and retention of study participants. | 12 Weeks

SECONDARY OUTCOMES:
Randomized participants complying with study visits and those lost to follow-up will be calculated.Compliance and follow-up are distinct because some participants may provide drinking patterns during follow-up regardless if they continue treatment. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: James C Garbutt, M.D., Principal Investigator — UNC-Chapel Hill